CLINICAL TRIAL: NCT02643017
Title: Effect of Dexmedetomidine on Postoperative Cognitive Function in Patients Undergoing Shoulder Arthroscopy With Beach Chair Position Under Desflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2015-0621
Record Dates: First submitted 2015-12-15; First posted 2015-12-30 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Rotator Cuff Tear
Keywords: cognitive function; desflurane; dexmedetomidine
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline
- Dex (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Administration of dexmedetomidine at a rate 0.6 ug/kg/hr during surgery.
  Arms: Dex
Drug: normal saline — Administration of same amount of dexmedetomidine at a rate 0.6 ug/kg/hr during surgery.
  Arms: normal saline

SUMMARY:
Investigate the effects of dexmedetomidine on postoperative cognitive function in patients undergoing shoulder arthroscopy with beach chair position under desflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing shoulder arthroscopic surgery with beach chair position

Exclusion Criteria:

1. Patients with respiratory disease
2. Patients with cardiac disease
3. Patients with cerebrovascular disease
4. patients with uncontrolled hypertension
5. Patients with dementia
6. Patients with psychiatric disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative cognitive decline assessed by mini-mental state examination | from 1 day before surgery to postoperative 1 day
  to compare cognitive decline after surgery between control and dexmedetomidine group with mini-mental state examination.
Number of patients with postoperative cognitive decline assessed by a battery of psychometric test | from 1 day before surgery to postoperative 1 day
  to compare cognitive decline after surgery between control and dexmedetomidine group with a battery of psychometric test. The battery consists of copy geometric form test, two-dimensional model test, grooved pegboard test, colored block design test, puzzle test, clock drawing test.

SECONDARY OUTCOMES:
Number of patients with increase of S100ß protein after surgery assessed by ELISA assay with blood of patients | from 5 min after induction of anesthesia to an 1 hour after surgery
  S100ß protein is the biologic marker for neuroinflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data.